CLINICAL TRIAL: NCT00667537
Title: A Phase I, Open-label, Dosimetry, Biodistribution and Pharmacokinetic Study of Alpharadin™ in Patients With Hormone Refractory Prostate Cancer and Skeletal Metastases
Brief Title: PK in Pts With HRPC & Skeletal Metastes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15302; 2006-006101-88 (EudraCT Number); BC1-05 (Other: Algeta ASA number)
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — radium Ra 223 dichloride; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radium-223 chloride (Experimental): IV administrations of 100 kBq/kg b.w (=110 kBq/kg based on the 2015 National Institute of Standards and Technology standardization). Two administrations took place with an interval of 6 weeks
  Interventions: Drug: Radium-223 chloride (Xofigo®, BAY88-8223) injection

INTERVENTIONS:
Drug: Radium-223 chloride (Xofigo®, BAY88-8223) injection — Sterile, clear and colourless aqueous solution of radium-223 chloride free of endotoxins, for intravenous administration

SUMMARY:
Primary objective: To investigate the biodistribution, radiation dosimetry, and pharmacokinetics of two separate intravenous (IV) injections of Xofigo (100 kBq/kg body weight [b.w.] [=110 kBq/kg based on the 2015 National Institute of Standards and Technology standardization], 6 weeks apart).

Secondary objectives: To determine the safety of IV injections of Xofigo after two separate injections (6 weeks apart), to evaluate treatment response (antitumour effect in osteoblastic bone metastases) of Xofigo treatment consisting of two injections of activity 100 kBq/kg b.w. (=110 kBq/kg based on the 2015 National Institute of Standards and Technology standardization), 6 weeks apart and to evaluate long term radiation toxicity and to collect survival data at 6 and 12 months after the first injection

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Hormone refractory with evidence of rising prostate-specific antigen (PSA): Subject must be maintained on androgen ablation therapy with luteinizing hormone-releasing hormone agonist or have undergone bilateral orchiectomy
* Serum testosterone level required to be ≤50 ng/dL
* Subjects who have received prior antiandrogen drug therapy: Flutamide, nilutamide, or cyproterone acetate must have stopped at least 4 weeks prior to study drug administration and progression, as defined by rising PSA as defined below, must have been demonstrated since cessation; bicalutamide must have stopped at least 6 weeks prior to study drug administration and progression, as defined by rising PSA as defined below, must have been demonstrated since cessation
* PSA progression: Progressive rise in PSA, defined as two consecutive increases in PSA documented over a previous reference value (measure 1). The first increase in PSA (measure 2) should occur at a minimum of 1 week from the reference value (measure 1). This increase in PSA should be confirmed (measure 3) after a minimum of 1 week. If the confirmatory PSA value (measure 3) is less than the previous value, the subject will still be eligible provided the next PSA measure (measure 4) is found to be greater than the second PSA value (measure 2)
* Skeletal metastases confirmed by bone scintigraphy within the last 6 weeks
* Performance status: Eastern Co-operative Oncology Group (ECOG) 0-2
* Life expectancy: ≥6 months
* Laboratory requirements: Neutrophil count ≥1.5 x 109/L, platelet count ≥100 x109/L, haemoglobin ≥95 g/L, total bilirubin level within normal institutional limits, aspartate aminotransferase and alanine aminotransferase ≤2.5 times upper institutional limit of the normal range, S Creatinine ≤1.5 times upper institutional limit of the normal range

Exclusion Criteria:

* Has received an investigational drug within 4 weeks prior to the administration of radium-223, or is scheduled to receive one during the treatment and post-treatment period
* Has received chemo-, immunotherapy, or external radiotherapy within the last 4 weeks prior to administration of study drug, or has not recovered from adverse events due to agents administered more than 4 weeks earlier
* More than one regimen of previous cytotoxic chemotherapy
* Has received prior hemibody external radiotherapy
* Has a need for immediate external radiotherapy
* Has received systemic radiotherapy with radium-223, strontium-89, samarium-153, rhenium-186 or rhenium-188 for the treatment of bony metastases within the last year prior to administration of study drug
* Has started treatment with bisphosphonates less than 3 months prior to administration of study drug. Patients are allowed to be on bisphosphonates provided patient is on a stable dose for >/= 12 weeks before administration of study drug
* Patients who are </= 4 weeks (6 weeks for bicalutamide) post withdrawal of antiandrogen therapy
* Patients who have started or stopped systemic steroids, within a week prior to study drug administration, or are expected to be subject to changes in the systemic steroid medication
* Other currently active (relapse within the last 3 years) malignancy (except non-melanoma skin cancer) that are not prostate cancer metastases
* Visceral (e.g. liver, lung) metastases from prostate cancer as assessed by abdominal/ pelvic CT or chest radiograph within six weeks before administration of study drug
* Lymph node metastases with short-axis diameter greater than 2 cm
* Bulky loco-regional disease
* Any other serious illness or medical condition, for example: any uncontrolled infection, any patient who has clinical heart failure severe enough to cause marked limitation of activity, and who is only comfortable at rest; or any patient who has heart failure more severe than this (NYHA Heart Failure Class III or IV), Crohns disease or ulcerative colitis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Estimation of whole-body retention of radioactivity at each imaging time post-injection | 1 week
Estimation of the individual organ uptake/retention of radioactivity at each time-point post injection | 1 week
Estimate retention of administered radioactivity in blood | Up to 1 week
Estimation of elimination of radioactivity in urine and faeces | 2 days
Calculation of estimated absorbed radiation dose to target organs | 1 week
Pharmacokinetics | 1 week

SECONDARY OUTCOMES:
Comparison of the biodistribution and dosimetry after the first and second injection | 7 weeks
Prostate specific antigen (PSA) response | At baseline, before injections, and at 2 month intervals during the 12 month follow up period
  PSA decline, defined as the number of patients with a confirmed ≥50% reduction in PSA level after treatment with respect to the pre-injection PSA level and the time to PSA progression after PSA response
Survival | 6 and 12 months after the first injection
Adverse events | 1 year
Laboratory variables; serum biochemistry and haematology | 1 year
Vital signs | 12 weeks
  Systolic/diastolic blood pressure, respiratory rate, heart rate and body temperature
ECG (12 leads) | 12 weeks
  Electrocardiogram (12 leads)
Physical examination | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Sutton, Surrey, United Kingdom

REFERENCES:
- [Result] Cook G Jr, Parker C, Chua S, Johnson B, Aksnes AK, Lewington VJ. 18F-fluoride PET: changes in uptake as a method to assess response in bone metastases from castrate-resistant prostate cancer patients treated with 223Ra-chloride (Alpharadin). EJNMMI Res. 2011 Jun 7;1(1):4. doi: 10.1186/2191-219X-1-4. PMID 22214491
- [Result] Chittenden SJ, Hindorf C, Parker CC, Lewington VJ, Pratt BE, Johnson B, Flux GD. A Phase 1, Open-Label Study of the Biodistribution, Pharmacokinetics, and Dosimetry of 223Ra-Dichloride in Patients with Hormone-Refractory Prostate Cancer and Skeletal Metastases. J Nucl Med. 2015 Sep;56(9):1304-9. doi: 10.2967/jnumed.115.157123. Epub 2015 Jul 16. PMID 26182965
- [Result] Hindorf C, Chittenden S, Aksnes AK, Parker C, Flux GD. Quantitative imaging of 223Ra-chloride (Alpharadin) for targeted alpha-emitting radionuclide therapy of bone metastases. Nucl Med Commun. 2012 Jul;33(7):726-32. doi: 10.1097/MNM.0b013e328353bb6e. PMID 22513884
- [Result] Hobbs RF, Song H, Watchman CJ, Bolch WE, Aksnes AK, Ramdahl T, Flux GD, Sgouros G. A bone marrow toxicity model for (2)(2)(3)Ra alpha-emitter radiopharmaceutical therapy. Phys Med Biol. 2012 May 21;57(10):3207-22. doi: 10.1088/0031-9155/57/10/3207. Epub 2012 May 1. PMID 22546715
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/